CLINICAL TRIAL: NCT04751357
Title: Argatroban Monitoring in Critically Ill Patients: Evaluation of a Novel Ecarin-based Bedside Test
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dr. Georg Scheriau, Principal investigator, Medical University of Vienna
Other Study IDs: EK Nr: 1635/2020
Record Dates: First submitted 2021-02-08; First posted 2021-02-12 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Heparin-induced Thrombocytopenia
Keywords: Argatroban; ECA-Test; Ecarin; Clot-Pro; Thrombelastometry; ROTEM

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: ECA-Test (Clot-Pro) — Thrombelastometric ECA-Test performed on Clot-Pro

SUMMARY:
Argatroban is a parenteral direct Thrombininhibitor used for anticoagulation in patients suffering from heparin induced thrombocytopenia (HIT). There is increasing evidence suggesting that the activated partial thromboplastine time (aPTT), which is recommended for dosage monitoring, correlates poorly with serum argatroban concentration in critically ill patients. Therefore it may be badly suited to determine the correct dosing. Ecarin based tests have been proven to be effective in determining effects of direct thrombin inhibitors. The investigators now plan to evaluate a novel, rotational thrombelastometric, ecarin based bedside test for its ability to measure the effect of argatroban in critically ill patients. So far an excellent correlation of a similar test could be shown in spiked plasma of healthy adults. According to the manufacturer the ECA-Test is able to detect direct thrombininhibitors. However to our knowledge neither the ECA-Test nor other ecarin-based thrombelastometric tests have been studied in critically ill patients treated with argatroban. The investigators therefore seek to investigate the correlation of the ECA-Test (ClotPro®) with the serum argatroban concentration.

ELIGIBILITY:
Inclusion Criteria:

* Continuous infusion of Argatroban in routine clinical use according to local standard of care
* Expected length of stay at ICU > 4 days
* 18 years

Exclusion Criteria:

* Heparin infusion in the last fourhours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients at the Intensive Care Unit who receive a continuous infusion of argatroban are eligible for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Correlation of ECA-Test CT with Argatroban Plasma Concentration | ECA-Test CT and Argatroban Plasma Concentration will be measured on five consecutive days starting with inclusion in the study on day 0.
  Correlation of ECA-Test CT with Argatroban Plasma Concentration on five consecutive days

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, General Hospital, Vienna, Austria